CLINICAL TRIAL: NCT06168617
Title: Feasibility Study of Tests, on the Model of Real-life Daily Tasks, Measuring the Performance of Different Vision Restoration Strategies, After Cataract Surgical Treatment With Different Types of Intraocular Lens Implants.
Brief Title: CAtaract ASSessment of IntrOcular Lens Objective PErformancE
Acronym: CASSIOPEE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier National d'Ophtalmologie des Quinze-Vingts (Other)
Collaborators: Fondation Ophtalmologique Adolphe de Rothschild (Network); StreetLab Vision (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: P22-08
Record Dates: First submitted 2023-12-01; First posted 2023-12-13 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Cataract
Keywords: Cataract; Intraocular Lens
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Intervention Model Description: Prospective, interventional, non-invasive, monocentric, longitudinal, non-randomized study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pilot phase (Experimental): 5 patients of both 3 groups will perform the parametric studying tasks. This phase aims at determine the feasibility of the tasks according to their parameters : Guided walk, visuo-manual task and posturography.
  Interventions: Diagnostic Test: Performance tasks in daily life
- Validation phase (Experimental): 20 patients of both 3 groups will perform these performance tasks. This phase is designed to evaluate the performance tests executed by patients in real-life situations.
  Interventions: Diagnostic Test: Performance tasks in daily life

INTERVENTIONS:
Diagnostic Test: Performance tasks in daily life — Evaluation of performance tests executed by patients in real-life situations.

SUMMARY:
Prospective, interventional, non-invasive, monocentric, longitudinal, non-randomized study

DETAILED DESCRIPTION:
There are many strategies for restoring vision after cataract surgery. They all involve the use of intraocular lenses (IOLs) to correct a single focal length (monofocal lenses) or several focal lengths (multifocal lenses). Each focal length corrected by the implants represents a distance of clear vision for patients. The complexity of the optical design and the neurosensory adaptation required for this restoration may present a downside, as implant patients may complain of light halos, glare or problems with depth perception, depending on the case.

Existing validated techniques are not sufficient to accurately assess the benefits or difficulties in the daily lives of elderly patients, the a With this project, the patient and his or her autonomy become the focus of the evaluation of IOL performance, particularly for IOLs of recent design, which makes it possible to better characterise the consequences of their implantation. PerfO studies of IOLs used in cataract surgery will be based on objectives tasks inspired by daily life performed by patients according to Street Lab procedures.

ELIGIBILITY:
Inclusion Criteria:

* Male / Female
* 65-75 years old
* Pseudophakia, implanted with 2 trifocal IOL or 2 EDOF IOL or with 2 monofocal IOL calculated for monovision
* Second eye surgery performed > 1 month before inclusion with stable residual refraction
* No degenerative or neurological disease
* Good understanding of the French language
* No use of an aid to locomotion (example: cane, etc...)
* Binocular far non corrected visual acuity ≥ 8/10
* Refraction at distance vision

  * Spherical equivalent in distance vision ≤ 0.75 diopter
  * Cylinder ≤ 0.75 diopter

Monovision group :

> Addition=1.25 diopter ±0.50

Multifocal group :

* Monocular far non corrected visual acuity ≥ 8/10
* ATLISA tri (Zeiss)

EDOF group :

* Monocular far non corrected visual acuity ≥ 8/10
* Eyehance (J&J)

Exclusion Criteria:

Media opacity or eye movement disorder (nystagmus) that interferes with retinal imaging data quality in the opinion of the investigator ;

* Media opacity or eye movement disorder (nystagmus) that interferes with retinal imaging data quality in the opinion of the investigator ;
* Any concurrent intraocular condition that, in the opinion of the investigator would either require surgical intervention during the study to prevent or treat visual loss that might result from that condition or affect interpretation of study results ;
* Known systemic illness which in the opinion of the investigator will prevent from actively participating in the study ;
* Concomitant treatment in either eye (concomitant use of vitamins/supplements is not excluded) ;
* Inability to comply with study task instructions or study visits ;
* Medication that may cause motor, visual or cognitive impairment (PSAs, neuroleptics, etc.) or interfere with study evaluations ;
* Other uncontrolled ophthalmic conditions that may interfere with study evaluation ;
* Participation in another clinical trial that may interfere with the present study ;
* Cognitive impairment, illiteracy, and subjects who do not speak the national language ;
* Paralysis may compromise ability to perform manual grasping tasks ;
* Pregnant or breastfeeding woman ;
* Patient under legal protection ("curatelle" or "tutelle") ;
* Patient denied freedom by a legal or administrative order.

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Locomotion - Guided walk | 3 months
  The operator measure the success and completion rates for daily life tests:
  The performance is measured with the walking speed and the foot placement precision. The walking balance is also evaluated by recording the pelvis position.
Static and dynamic posturography with optical flow: | 3 months
  Postural control will be described by the Root Mean Square (RMS) of body sway in sagittal and coronal plans, the path length of the projection of the center of mass (CoM), the sway area described by the confidence ellipse which is the region that contains 95% of all COM samples. To better understand the visual, vestibular and somatosensory contributions on postural control, Romberg quotient (QR), Visual ratio (ViR), vestibular ratio (VeR) and somatosensory ratio (SR) will be calculated thanks to sensory conditions. Correlations with visual functions will be realized and postural deficits will be integrated into the locomotion score as a covariable.
Visuo-manual task | 3 months
  The variables analyzed :the duration of the visual search, which will be an indicator of the quality and ease of vision ; the duration of the grasping movement, which will be an indicator of the ease of the approach movement towards a low contrast object ; the duration between the seizure of the object and its deposit, which will be an indicator of the sensitivity to contrast ; the number of errors (wrong object grasped, object dropped, ...), will be an indicator of insufficient vision to perform the task.
Quality of life | 3 months
  French version Adapted Catquest-9SF questionnaire. It is a psychometric questionnaire specifically designed for cataracts. It assesses patient satisfaction with their eyesight. It consists of nine questions divided into two parts. The first part concerns two questions on the general quality of vision perceived by the patient, and the second part concerns seven questions on the difficulties that vision can cause on daily activities. The first page contains an explanatory note on the questionnaire. The patients' answers are divided into four equal boxes designating the degree of difficulty: very great difficulty, great difficulty, moderate difficulty and no difficulty.

CONTACTS AND LOCATIONS:
Overall Officials: Anna GEMAHLING, Principal Investigator — Fondation Hôpital Adolphe de Rothschild; Erci GABISON, Study Director — Fondation Hôpital Adolphe de Rothschild